CLINICAL TRIAL: NCT01005043
Title: Phase I/II Therapy Trial to Determine the Safety and Efficacy of Heavy Ion Radiotherapy in Patients With Osteosarcoma
Brief Title: Therapy Trial to Determine the Safety and Efficacy of Heavy Ion Radiotherapy in Patients With Osteosarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Dietmar Hopp Stiftung (Other)
Responsible Party: Principal Investigator, Juergen Debus, Prof. Dr. Dr. Jürgen Debus, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HITHD-01
Record Dates: First submitted 2009-10-23; First posted 2009-10-30 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Osteosarcoma
Keywords: non-resectable osteosarcoma; heavy ion radiotherapy; particle therapy; safety; toxicity; survival; radiotherapy
MeSH Terms: conditions — Osteosarcoma | interventions — Heavy Ion Radiotherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- heavy ion radiotherapy (Experimental): Heavy ion radiotherapy of osteosarcoma with 60 to 66 GyE (20-22 days). Before and after radiotherapy, but not during radiotherapy, chemotherapy is recommended to standard therapy protocols like EURAMOS 1 which is not part of this study.
  Interventions: Radiation: heavy ion radiotherapy (C12)

INTERVENTIONS:
Radiation: heavy ion radiotherapy (C12) — Desired target of Heavy ion radiotherapy is 60 to 66 Cobalt Gray Equivalent (GyE), whenever possible. It is applied through 1 - 3 isocenter treatment portals. Dose distributions are calculated and dose volume histograms (DVH) are generated. A α/β-ratio of 2 is used for biological plan optimization. Fractionation is planned to be equivalent to 6 x 3 GyE / week. Dosage to organs at risk is minimized. Treatment continues for 20 to 22 days or until one of the following criteria applies:
  Other illness that prevents further administration of treatment, Patient or legal guardian decides to withdraw from the study, or changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.
  Other Names: Particle therapy; Radiotherapy with C12; Ion therapy

SUMMARY:
The primary objectives of this trial are the determination of feasibility and toxicity of Heavy Ion Radiotherapy (C12) in patients with non-resectable osteosarcoma. Secondary endpoints are tumor response, disease free survival and overall survival. The aim is to improve outcome for patients with non-resectable osteosarcoma.

DETAILED DESCRIPTION:
Osteosarcoma is the most common primary malignant bone tumor in children and adolescents. For effective treatment, local control of the tumor is absolutely critical, because the chances of long term survival are <10% and might effectively approach zero if a complete surgical resection of the tumor is not possible. Up to date there is no curative treatment protocol for patients with non-resectable osteosarcomas, who are excluded from current osteosarcoma trials , e.g. EURAMOS1. Local photon radiotherapy has previously been used in small series and in an uncontrolled, highly individualized fashion, which, however, documented that high dose radiotherapy can, in principle, be used to achieve local control. Generally the radiation dose that is necessary for a curative approach can hardly be achieved with conventional photon radiotherapy in patients with non-resectable tumors that are usually located near radiosensitive critical organs such as the brain, the spine or the pelvis. In these cases Heavy Ion Radiotherapy (HIT) may offer a promising new alternative. Moreover, compared with photons, heavy ion particles provide a higher physical selectivity because of their finite depth coverage in tissue. They achieve a higher relative biological effectiveness. Phase I/II dose escalation studies of HIT in adults with non-resectable bone and soft tissue sarcomas have already shown favorable results.

Methods/Design: This is a monocenter, non-randomized study for patients older than 6 years of age with non-resectable osteosarcoma. Desired target dose is 60-66 Cobalt Gray Equivalent (GyE). Weekly fractionation of 6 x 3 Gy E is used. HIT will be administered exclusively at the Ion Radiotherapy Center in Heidelberg. Furthermore, FDG-PET imaging characteristics of non-resectable osteosarcoma before and after HIT will be investigated prospectively. Systemic disease before and after HIT is targeted by standard chemotherapy protocols and is not part of this trial.

The primary objectives of this trial are the determination of feasibility and toxicity of HIT. Secondary endpoints are tumor response, disease free survival and overall survival. The aim is to improve outcome for patients with non-resectable osteosarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of high grade osteosarcoma with or without metastases
* Non-resectable tumor of the pelvis, the skull base or the spine, respectively, incomplete or intralesional tumor resection - as confirmed after evaluation by two orthopedic surgeons (respectively neurosurgeons in case of spine tumors): one local surgeon and one referee surgeon of the University of Heidelberg.
* Age older than 6 years before start of radiotherapy
* Adequate performance status (Karnofsky >60%)
* Adequate blood cell production before the start of HIT in patients with pelvic or spine tumors as defined by: total white cell count (WBC) >1,0/nl; neutrophils > 200/µl; platelet count >20/nl
* No febrile neutropenia (neutrophils < 200/µl)
* Written informed consent of the patient or the legal guardians

Non-resectable tumor site means primary tumors affecting anatomic areas of the human body where a surgical total resection (R0) of the tumor is not possible for technical reasons, for example osteosarcoma of the pelvis, spine or the skull base. In any other cases, surgical resection is recommended.

Non-resectability has to be confirmed after evaluation by two orthopedic surgeons (respectively neurosurgeons in case of spine tumors): one local surgeon and one referee surgeon of the University of Heidelberg.

In some cases surgery of the tumor might be possible after HIT. Then we recommend surgical resection of residual tumor afterwards.

Exclusion Criteria:

* Age younger than 6 years
* Previous radiotherapy of the field that has to be radiated now
* Implanted metal within the planned radiation field, that leads to significant artefacts within the target volume
* Patients receiving any other investigational agents during the time of HIT
* Performance status (Karnofsky) < 60%)
* Pregnancy
* No written informed consent of patient or the legal guardians

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
feasibility, toxicity (tox) measured by the CTC Criteria .Unacceptable:grade 4 tox. A rate of acute tox (≤ 3 months during/after RT) > grade 3 of ≤ 5% and a rate of late tox > grade 3 of ≤ 3% will be acceptable. | before, weekly during RT and at follow-up (1, 6 and 19 weeks, 6, 12, 24, 36 48 and 60 months after RT).

SECONDARY OUTCOMES:
tumor response (RECIST criteria), disease free survival, overall survival and description of FDG-PET characteristics before and after RT. | 6, 12, 24, 36 48 and 60 months after RT

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, Head of Dep., Principal Investigator — Heidelberger Ionenstrahltherapiezentrum, HIT, Im Neuenheimer Feld 400, 69120 Heidelberg, Germany
Locations (1):
- Heidelberger Ionenstrahltherapiezentrum (HIT), Im Neuenheimer Feld 400, Heidelberg, Germany

REFERENCES:
- [Background] Bielack SS, Wulff B, Delling G, Gobel U, Kotz R, Ritter J, Winkler K. Osteosarcoma of the trunk treated by multimodal therapy: experience of the Cooperative Osteosarcoma study group (COSS). Med Pediatr Oncol. 1995 Jan;24(1):6-12. doi: 10.1002/mpo.2950240103. PMID 7968796
- [Background] Kamada T, Tsujii H, Tsuji H, Yanagi T, Mizoe JE, Miyamoto T, Kato H, Yamada S, Morita S, Yoshikawa K, Kandatsu S, Tateishi A; Working Group for the Bone and Soft Tissue Sarcomas. Efficacy and safety of carbon ion radiotherapy in bone and soft tissue sarcomas. J Clin Oncol. 2002 Nov 15;20(22):4466-71. doi: 10.1200/JCO.2002.10.050. PMID 12431970
- [Background] Oya N, Kokubo M, Mizowaki T, Shibamoto Y, Nagata Y, Sasai K, Nishimura Y, Tsuboyama T, Toguchida J, Nakamura T, Hiraoka M. Definitive intraoperative very high-dose radiotherapy for localized osteosarcoma in the extremities. Int J Radiat Oncol Biol Phys. 2001 Sep 1;51(1):87-93. doi: 10.1016/s0360-3016(01)01603-0. PMID 11516856
- [Background] Zhang H, Yoshikawa K, Tamura K, Tomemori T, Sagou K, Tian M, Kandatsu S, Kamada T, Tsuji H, Suhara T, Suzuki K, Tanada S, Tsujii H. [(11)C]methionine positron emission tomography and survival in patients with bone and soft tissue sarcomas treated by carbon ion radiotherapy. Clin Cancer Res. 2004 Mar 1;10(5):1764-72. doi: 10.1158/1078-0432.ccr-0190-3. PMID 15014030
- [Derived] Blattmann C, Oertel S, Schulz-Ertner D, Rieken S, Haufe S, Ewerbeck V, Unterberg A, Karapanagiotou-Schenkel I, Combs SE, Nikoghosyan A, Bischof M, Jakel O, Huber P, Kulozik AE, Debus J. Non-randomized therapy trial to determine the safety and efficacy of heavy ion radiotherapy in patients with non-resectable osteosarcoma. BMC Cancer. 2010 Mar 12;10:96. doi: 10.1186/1471-2407-10-96. PMID 20226028